CLINICAL TRIAL: NCT06818227
Title: MonPsyMoi: Etude Des Conditions d'implémentation et de l'Impact de la Plateforme Digitale française de Recueil de l'expérience Patient en Psychiatrie (Modules Avec et Sans " Feedback ")
Brief Title: MonPsy&Moi: A Digital Platform for Collecting Patient-Reported Experience and Outcome Measures in Psychiatry
Acronym: Mon Psy & Moi
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: RCAPHM21_0429
Record Dates: First submitted 2025-01-27; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Schizophrenia Disorders; Bipolar Disorders; Major Depression
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Psychiatric patients

SUMMARY:
Mental health disorders, with a 30% annual prevalence rate, are a leading cause of disability and reduced life expectancy. Despite their impact, patient-reported experience measures (PREMs) and outcome measures (PROMs) are underutilized in psychiatry. MonPsy&Moi®, a digital platform funded by ATIH and DGOS, addresses this gap by providing a user-friendly tool to assess patient experiences and outcomes in real-time, aiming to improve the quality of psychiatric care across France.

The study consists of two stages:

Stage 1 (No Feedback): MonPsy&Moi® is deployed across 12 psychiatric facilities, collecting patient data without feedback to clinicians. Objectives include assessing implementation feasibility, validating adaptive questionnaires (PREMIUM), and identifying predictors of patient outcomes, such as relapse and healthcare utilization.

Stage 2 (With Feedback): Focuses on patients with severe mental illnesses (schizophrenia, bipolar disorders, and major depressive disorders). This stage evaluates the impact of providing PREMs/PROMs feedback to clinicians on relapse rates, healthcare costs, and overall patient outcomes.

MonPsy&Moi® uses adaptive questionnaires tailored to psychiatric care, covering key domains such as dignity, information, interpersonal relationships, care environment, and treatment. It also evaluates health-related quality of life, including psychological well-being, autonomy, self-esteem, and social relationships. The platform integrates with national healthcare databases (SNDS) to enhance data analysis and predict patient trajectories.

The study will involve over 22,000 participants in Stage 1 and 1,100 participants in Stage 2, using a quasi-experimental design to compare feedback and non-feedback strategies. Results aim to demonstrate the feasibility, acceptability, and efficacy of MonPsy&Moi® in improving mental health outcomes and guiding national psychiatric care policies.

By empowering patients and clinicians with actionable insights, MonPsy&Moi® aspires to set a new standard for patient-centered mental healthcare in real-world settings

ELIGIBILITY:
Inclusion Criteria:

* Residing in France. Age between 18 and 65 years at the time of inclusion.

Receiving care in one of the 12 participating psychiatric facilities, with a confirmed diagnosis of:

Schizophrenia Spectrum Disorders (e.g., schizophrenia, schizoaffective disorder).

Bipolar Disorders. Major Depressive Disorders. A valid email address. Ability to read and understand French. Non-opposition to participating in the study (based on informed consent).

Exclusion Criteria:

* Primary diagnosis of an organic mental disorder, including:

Dementia. Stroke. Traumatic brain injury. Individuals deprived of liberty by judicial decision (e.g., incarcerated patients).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adults residing in France and receiving care in 12 participating psychiatric facilities. The focus is on adults aged 18-65 with severe mental illnesses, such as schizophrenia spectrum disorders, bipolar disorders, and major depressive disorders. Participants must have a valid email address, understand French, and not oppose participation. Vulnerable populations, such as those under involuntary psychiatric care, are included to assess care quality, while individuals with organic mental disorders or those deprived of liberty are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 23660 (Estimated)
Dates: Start 2025-02-02 (Estimated); Primary Completion 2026-09-21 (Estimated); Study Completion 2026-09-21 (Estimated)

PRIMARY OUTCOMES:
Relapse at 12 Months | within 12 months
  Relapse is defined as one or more of the following events occurring within 12 months:Full-time psychiatric hospitalization, Psychiatric emergency care.
  Hospitalization due to a suicide attempt, Death.

SECONDARY OUTCOMES:
Impact of Feedback on healthcare resource utilization | 6 and 12 months post-inclusion
  Mortality at 6 and 12 months.
Cost-Effectiveness Analysis | 12 months post-inclusion
  Incremental cost-effectiveness ratio (ICER) and cost-utility analysis (cost per relapse avoided or per quality-adjusted life year [QALY] gained).

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No